CLINICAL TRIAL: NCT00825201
Title: Phase I Trial of Intraperitoneal Nab-Paclitaxel (Abraxane) in the Treatment of Advanced Malignancies Primarily Confined to the Peritoneal Cavity
Brief Title: Intraperitoneal Paclitaxel Albumin-Stabilized Nanoparticle Formulation in Treating Patients With Advanced Cancer of the Peritoneal Cavity
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); National Comprehensive Cancer Network (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 08059; CHNMC-08059; ABRAXIS-CHNMC-08059; NCCN-A02; CDR0000632797 (Registry Identifier: NCI PDQ); NCI-2010-00921 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2009-01-16; First posted 2009-01-19 (Estimated); Last update posted 2018-01-19 (Actual); Status verified 2018-01

CONDITIONS: Ovarian Cancer; Peritoneal Cavity Cancer; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: peritoneal carcinomatosis; peritoneal cavity cancer; stage IV ovarian epithelial cancer; recurrent ovarian epithelial cancer; unspecified adult solid tumor, protocol specific
MeSH Terms: conditions — Ovarian Neoplasms; Peritoneal Neoplasms; Carcinoma, Ovarian Epithelial | interventions — Taxes; Albumin-Bound Paclitaxel; 130-nm albumin-bound paclitaxel; Chromatography, Liquid; Mass Spectrometry

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (paclitaxel albumin-stabilized nanoparticle) (Experimental): Patients receive paclitaxel albumin-stabilized nanoparticle formulation given IP on days 1, 8, and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: paclitaxel albumin-stabilized nanoparticle formulation; Other: liquid chromatography; Other: mass spectrometry; Other: pharmacological study; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: paclitaxel albumin-stabilized nanoparticle formulation — Given IP
  Other Names: ABI-007; nab paclitaxel; nab-paclitaxel; nanoparticle albumin-bound paclitaxel
Other: liquid chromatography — Plasma and peritoneal fluid samples will be collected prior to nab-paclitaxel, at completion of nab-paclitaxel infusion and at hours 1, 2, 4, 6, 8, 12, 24 and 48 following completion of infusion.
Other: mass spectrometry — Plasma and peritoneal fluid samples will be collected prior to nab-paclitaxel, at completion of nab-paclitaxel infusion and at hours 1, 2, 4, 6, 8, 12, 24 and 48 following completion of infusion.
Other: pharmacological study — Plasma and peritoneal fluid samples will be collected prior to nab-paclitaxel, at completion of nab-paclitaxel infusion and at hours 1, 2, 4, 6, 8, 12, 24 and 48 following completion of infusion.
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as paclitaxel albumin-stabilized nanoparticle formulation, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving paclitaxel albumin-stabilized nanoparticle formulation directly into the abdomen may kill more tumor cells.

PURPOSE: This phase I trial is studying the side effects and best dose of intraperitoneal paclitaxel albumin-stabilized nanoparticle formulation in treating patients with advanced cancer of the peritoneal cavity.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES: I. To determine the maximally tolerated dose (MTD) of nab-paclitaxel as a single agent administered intraperitoneally via an intraperitoneal catheter.

SECONDARY OBJECTIVES: I. To evaluate the pharmacokinetics of nab-paclitaxel (Abraxane) in the plasma and peritoneum when it is administered directly into the peritoneal cavity. II. To determine the potential pharmacokinetic advantage (favorable ratio of nab-paclitaxel (Abraxane) concentration in the peritoneal cavity vs. plasma) for nab-paclitaxel administered intraperitoneally. III. To determine the progression of peripheral neuropathy in patients treated with intraperitoneal chemotherapy on this study through pre-treatment and sequential evaluation of the Neuropathic Pain Syndrome Inventory and Serial Nerve Conduction Studies.

OUTLINE: This is a dose-escalation study. Patients receive paclitaxel albumin-stabilized nanoparticle formulation given intraperitoneally (IP) on days 1, 8, and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histological confirmed advanced cancer primarily confined to the peritoneal cavity which have progressed on previous chemotherapeutic regimens, or for which no "standard" chemotherapeutic regimens exist
* Prior taxane exposure is allowed; prior IP chemotherapy is allowed, if it was not complicated by peritoneal adhesions; patients with ovarian cancer having residual disease at second-look laparotomy or following secondary debulking are also eligible; patients must be 4-6 weeks after surgery and they must have recovered from the surgery prior to initiating IP chemotherapy
* Eastern Cooperative Oncology Group (ECOG) less than or equal to 2
* Life expectancy of greater than 3 months
* Absolute neutrophil count > 1,500/mcL
* Platelets > 100,000/mcL
* Total bilirubin within normal institutional limits
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamic pyruvic transaminase [SGPT]) < 2.5 x institutional upper limit of normal
* Creatinine within normal institutional limits or creatinine clearance > 60 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal
* Documentation of measurable disease (with baseline measurements taken with 4 weeks of study entry, when present and appropriate); presence of measurable disease is not, per se, a prerequisite for entry onto this study
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administer more than 4 weeks earlier; there is no limit on the number of prior lines of chemotherapy
* Patients may not be receiving any other investigational agents
* Patients with known brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to nab-paclitaxel
* Patients with ongoing abdominal infections or bowel obstruction
* Patients with known peritoneal adhesions that preclude the placement of an intraperitoneal catheter in the opinion of the surgeon placing the intraperitoneal catheter
* Pre-existing grade >= 2 sensory neuropathy
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study; breastfeeding should be discontinued if the mother is treated with nab-paclitaxel
* Human immunodeficiency virus (HIV)-positive patients on combination antiretroviral therapy
* "Massive Ascites" requiring therapeutic paracentesis, will not be cause for ineligibility, per se, it will be evaluated on an individual basis; investigators who have any questions regarding assessing ascites are asked to speak with the Principal Investigator

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2009-01; Primary Completion 2018-01-16 (Actual); Study Completion 2018-01-16 (Actual)

PRIMARY OUTCOMES:
Dose-limiting toxicities as assessed by Common Terminology Criteria for Adverse Events (CTCAE) version 3.0 and maximum-tolerated dose | 28 days following the first course of treatment in which 2 or more patients experience a Dose Limiting Toxicity
  The toxicities observed at each dose level will be summarized in terms of type (organ affected or laboratory determination such as absolute neutrophil count), severity (by CTCAE and nadir or maximum values for the laboratory measures), time of onset (i.e., course number), duration, and reversibility or outcome. Tables will be created to summarize these toxicities and side effects by dose and course.

SECONDARY OUTCOMES:
Response according to Response Evaluation Criteria in Solid Tumors (RECIST) | 4 weeks after completion of the last course of treatment
  All responses will be reported; because of the potential heterogeneity of the patients, no attempt will be made to estimate the response rate.

OTHER OUTCOMES:
Pharmacokinetic (area under the curve [AUC], pharmacological advantage, and clearance in the plasma and peritoneum) | Course 1 days 1 and 15 at 1, 2, 4, 6, 8, 12, 24, and 48 hours
  Will be summarized by dose level with simple summary statistics: means (possibly after transformation) or medians, ranges, and standard deviations (if numbers and distribution permit).
Pharmacodynamic (AUC, pharmacological advantage, and clearance in the plasma and peritoneum) | Course 1 days 1 and 15 at 1, 2, 4, 8, 12, 24 and 48 hours
  Will be summarized by dose level with simple summary statistics: means (possibly after transformation) or medians, ranges, and standard deviations (if numbers and distribution permit).

CONTACTS AND LOCATIONS:
Overall Officials: Mihaela Cristea, MD, Principal Investigator — City of Hope Comprehensive Cancer Center; Mihaela Cristea, MD, Study Chair — City of Hope Comprehensive Cancer Center
Locations (2):
- United States (2):
  - City of Hope Medical Center, Duarte, California
  - Swedish Medical Center, Seattle, Washington

REFERENCES:
- [Derived] Cristea MC, Frankel P, Synold T, Rivkin S, Lim D, Chung V, Chao J, Wakabayashi M, Paz B, Han E, Lin P, Leong L, Hakim A, Carroll M, Prakash N, Dellinger T, Park M, Morgan RJ. A phase I trial of intraperitoneal nab-paclitaxel in the treatment of advanced malignancies primarily confined to the peritoneal cavity. Cancer Chemother Pharmacol. 2019 Mar;83(3):589-598. doi: 10.1007/s00280-019-03767-9. Epub 2019 Jan 8. PMID 30623229